CLINICAL TRIAL: NCT02130557
Title: A MULTICENTER PHASE 3 RANDOMIZED, OPEN-LABEL STUDY OF BOSUTINIB VERSUS IMATINIB IN ADULT PATIENTS WITH NEWLY DIAGNOSED CHRONIC PHASE CHRONIC MYELOGENOUS LEUKEMIA
Brief Title: A Multicenter Phase 3, Open-Label Study of Bosutinib Versus Imatinib in Adult Patients With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV001; 2013-005101-31 (EudraCT Number); B1871053 (Other: Alias Study Number)
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Leukemia, Myelogenous, Chronic, Breakpoint Cluster Region-Abelson Proto-oncogene (BCR-ABL) Positive
Keywords: Leukemia; Myelogenous; Chronic; BCR-ABL Positive; Bosutinib; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome; Neoplasms by Histologic Type; Bone Marrow Diseases; Hematologic Diseases; Translocation, Genetic; Pathologic Processes; Imatinib; Therapeutic Uses; Pharmacologic Actions; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome; Neoplasms by Histologic Type; Bone Marrow Diseases; Hematologic Diseases; Translocation, Genetic; Pathologic Processes | interventions — bosutinib; Imatinib Mesylate

STUDY DESIGN:
Masking Description: NOTE: Value was Open Label in old format; This study has an open-label design. Although most efficacy studies have a double blind design, this is not feasible in this trial, due to the complexity of the dose reduction and dose escalation schemes with tablets of various sizes, dosage strengths, as well as the number of tablets that would be required daily. However, the opportunity for bias is mitigated by the use of objective outcome measures (MMR, CCyR, CHR). The Investigators will be instructed to ensure that laboratory/pathology personnel are blinded to treatment information. For these reasons, an open-label, randomized study is appropriate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bosutinib (Experimental): Bosutinib, 400 mg, oral administration once a day
  Interventions: Drug: Bosutinib
- Imatinib (Active Comparator): Imatinib, 400 mg, oral administration once a day
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Bosutinib — Bosutinib (Bosulif®) is an orally bioavailable, potent, multi-targeted, dual Src-Abl tyrosine kinase inhibitor (TKI) that has been approved for the treatment of adult patients with Philadelphia positive (Ph+) chronic phase (CP), accelerated phase (AP) and blast phase (BP) chronic myelogenous leukemia (CML) previously treated with other TKI inhibitor therapy.[1] This study will investigate the use of bosutinib as first-line treatment for patients with Ph+ CP CML.
  Arms: Bosutinib
Drug: Imatinib — Imatinib mesylate (referred to in this protocol as imatinib) is an inhibitor of the BCR-ABL kinase and been the standard first-line therapy for patients with chronic-phase CML. Imatinib was granted approval by the European Commission in November 2001 and by the FDA in December 2002 for the treatment of newly diagnosed patients with CP Ph+ CML based on results from the IRIS trial.
  Imatinib is considered the standard of care for both first-line and later line settings, and consequently is an appropriate active comparator.
  Arms: Imatinib

SUMMARY:
Phase 3, 2-arm, randomized, open label trial. Patients will be randomized to receive bosutinib or imatinib for the duration of the study.

DETAILED DESCRIPTION:
The study will be open for enrollment until the planned number of approximately 500 Philadelphia Chromosome Positive (Ph+) patients have been randomized (approximately 250 Ph+ patients in each treatment arm; a total of approximately 530 Ph+ and Ph- patients). All patients will be treated and/or followed for approximately 5 years (240 weeks) after randomization until the study has closed. Patients who discontinue study therapy early due to disease progression or intolerance to study medication will continue to be followed yearly for survival for up to approximately 5 years (240 weeks) after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Molecular diagnosis of CP CML of ≤ 6 months (from initial diagnosis).
2. Adequate hepatic, renal and pancreatic function.
3. Age ≥ 18 years.

Exclusion Criteria:

1. Any prior medical treatment for CML, including tyrosine kinase inhibitors (TKIs), with the exception of hydroxyurea and/or anagrelide treatment, which are permitted for up to 6 months prior to study entry (signature of ICF) if suitably approved for use in the subject's region.
2. Any past or current Central Nervous System (CNS) involvement, including leptomeningeal leukemia.
3. Extramedullary disease only.
4. Major surgery or radiotherapy within 14 days of randomization.
5. History of clinically significant or uncontrolled cardiac disease.
6. Known seropositivity to human immunodeficiency virus (HIV), current acute or chronic hepatitis B (hepatitis B surface-antigen positive), hepatitis C, cirrhosis or evidence of decompensated liver disease. Patients with resolved Hepatitis B can be included.
7. Recent or ongoing clinically significant GI disorder, e.g. Crohn's Disease, Ulcerative Colitis, or prior total or partial gastrectomy.
8. History of another malignancy within 5 years with the exception of basal cell carcinoma or cervical carcinoma in situ or stage 1 or 2 cancer that is considered adequately treated and currently in complete remission for at least l2 months.
9. Current, or recent (within 30 days, or 5 half-lives of investigational product) participation in other clinical trials of investigational agents and/or containing interventional procedures deemed contrary to the objectives and conduct of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2020-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (188):
- United States (64):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - Saint Alphonsus Regional Medical Center, Cancer Care Center, Boise, Idaho
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Alphonsus Caldwell Cancer Care Center, Caldwell, Idaho
  - Saint Alphonsus Medical Center Nampa, Nampa, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - PHARMACY Department Franciscan St. Francis Health ATTN:Jill Leslie, Pharm D, Indianapolis, Indiana
  - Cancer Center of Acadiana at Lafayette General Medical Center, Lafayette, Louisiana
  - Lafayette General Medical Center, Lafayette, Louisiana
  - LSU Health Sciences Center-Shreveport, Shreveport, Louisiana
  - University Health Shreveport, Shreveport, Louisiana
  - Rcca Md Llc, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, ONC/Research Pharmacy, Worcester, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St. Joseph Mercy Hospital - Inpatient Pharmacy, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - St. Joseph Mercy-Brighton, Brighton, Michigan
  - St. Joseph Mercy-Canton, Canton, Michigan
  - Chelsea Community Hospital, Chelsea, Michigan
  - St. John Hospital&Medical Center, Detroit, Michigan
  - St. John Hospital&Medical Center-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Van Elslander Cancer Center, Pharmacy, Grosse Pointe Woods, Michigan
  - Minnesota Oncology Hematology, PA, Edina, Minnesota
  - Park Nicollet Frauenshuh Cancer center, Saint Louis Park, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - North Mississippi Medical Center Hematology and Oncology Clinic, Tupelo, Mississippi
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - NYU Winthrop Hospital - Oncology / Hematology department, Mineola, New York
  - NYU Winthrop Hospital - Pharmacy Department, Mineola, New York
  - Beth Israel Medical Center, New York, New York
  - University of Rochester Investigational Drug Pharmacy, Rochester, New York
  - University of Rochester, Rochester, New York
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UC Health Physicians Office South,, West Chester, Ohio
  - MUSC University Hospital, Charleston, South Carolina
  - MUSC University of South Carolina, Investigational Drug Services, Charleston, South Carolina
  - MUSC-Hollings Cancer Center, Charleston, South Carolina
  - GHS Cancer Institute, Easley, South Carolina
  - GHS Cancer Institute, Greenville, South Carolina
  - GHS Cancer Institute, Greer, South Carolina
  - GHS Cancer Institute, Seneca, South Carolina
  - GHS Cancer Institute, Spartanburg, South Carolina
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Murray, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - HSHS St. Vincent Hospital Regional Cancer Center at HSHS St. Vincent Hospital, Green Bay, Wisconsin
  - HSHS St. Vincent Hospital, Green Bay, Wisconsin
  - HSHS St. Vincent Hospital Regional Cancer Center at HSHS St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - St George Hospital - Hematology Department, Kogarah, New South Wales
  - Eastern Clinical Research Unit, Level 2, Box Hill, Victoria
- Belgium (4):
  - UZ Ghent (University Hospital Ghent), Ghent
  - Department of Haematology at UZ Leuven (7 th Floor), Leuven
  - Hematology Department of CHU de Liège, Liège
  - Hematology Department CHR Verviers, Verviers
- Canada (7):
  - Horizon Health Network - The Moncton Hospital, Moncton, New Brunswick
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Québec - Université Laval, Québec
- Czechia (4):
  - Fakultní Nemocnice Brno, Brno
  - Fakultní Nemocnice Hradec Králové, Hradec Králové
  - Fakultní nemocnice Olomouc, Olomouc
  - Všeobecná fakultní Nemocnice v Praze, Prague
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Roskilde Hospital, Roskilde
- Helsinki University Central Hospital, Helsinki, Finland
- France (9):
  - Oncologie Centre de Radiotherapie, Strasbourg, NC
  - Institut Bergonié, Bordeaux
  - private Practice of Pr Philippe Rousselot, Le Chesnay
  - private Practice of Dr. Viviane Dubruille, Nantes
  - Hôpital L'Archet 1-CHU Nice, Nice
  - Institut de Cancérologie du Gard - Hématologie Clinique, Nîmes
  - Pr Mauricette Michallet Centre Hospitalier Lyon Sud, Pierre-Bénite
  - INSERM CIC 1402 - CHU Poitiers, Poitiers
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
- Germany (7):
  - Universitätsklinikum Bonn, Bonn, Rhineland-Palatinate
  - Uniklinikum Aachen, Aachen
  - Charité, CVK, Med. Klinik m.S Hämatologie und Onkologie, Berlin
  - Universitätsklinikum Freiburg, Klinik für Innere Medizin I, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Onkologisches Zentrum, Hamburg
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Jena Lobeda-Ost
  - Schwerpunktpraxis für Hämatologie und Onkologie, Magdeburg
- Hungary (6):
  - Semmelweis Egyetem I. Belgyógyászat, Budapest
  - Debreceni Egyetem Klinikai Központ, Belgyógyászati Inézet Hematológiai Tanszék, Debrecen
  - Petz Aladár Megyei OktatóKórház, II. Belgyógyászati Osztály és Haematológiai Részleg, Győr
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Szegedi Tudományegyetem, AOK, Szent-Györgyi Albert Klinikai Központ, II. sz., Szeged
  - Jász-Nagykun-Szolnok Megyei Hetényi, Géza Kórház-Rendelőintézet, Szolnok
- Israel (2):
  - Hematology Department, Rambam Medical Centre, Haifa
  - Hematology Div. Davidoff Cancer Center, Rabin Medical Center, Petah Tikva
- Italy (11):
  - Azienda Ospedaliero-Universitaria "Policlinico - Vittorio Emanuele" - P.O. G. Rodolico, Catania, CT
  - USC Ematologia, A. O. Papa Giovanni XXIII, Bergamo
  - Policlinico S. Orsola - Malpighi,, Bologna
  - A.O. Brozu - P.O. Armando Businco, Cagliari
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - IRCCS - AOU San Martino_IST, Ematologia 1, Genova
  - Istituto Scientifico San Raffaele, Milan
  - Unità di Ricerca Clinica, U.O. Ematologia Adulti, Monza
  - A.O.U. Policlinico Università degli Studi di Napoli "Federico II", Napoli
  - Dipartimento di ematologia, Reggio Calabria
  - ASL Roma 2 - Ospedale Sant'Eugenio, Roma
- Mexico (2):
  - Hospital Angeles del Pedregal (S.A. de C.V.), Mexico City, Mexico City
  - Monterrey International Research Center, Monterrey, Nuevo León
- Netherlands (2):
  - Klinische Farrnacologie en Apotheek, Amsterdam, North Holland
  - VU University Medical Center, Amsterdam, North Holland
- Norway (2):
  - Haukeland University Hospital Department of Hematology, Bergen
  - St. Olavs Hospital, Trondheim
- Poland (7):
  - Klinika Hematologii i Transplantologii Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - SPZOZ ZSM w Chorzowie Oddzial Hematologiczny, Chorzów
  - Samodzielny Publiczny Szpital Kliniczny im. A Mielęckiego, ŚUM w Katowicach, Katowice
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Hematologii, Krakow
  - Wojewódzki Szpital Specjalistyczny im M. Kopernika, Klinika Hematologii Uniwersytetu Medycznego, Lodz
  - SPSK, Klinika Hematoonkologii i Transplantacji Szpiku w Lublinie, Lublin
  - Universytet Medyczny im. Piastów Śląskich we Wrocławiu Katedra i, Wroclaw
- Singapore (3):
  - National University Hospital, Main Building, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Univerzitná Nemocnica Bratislava-Nemocnica sv. Cyrila a Metoda, Bratislava, Slovakia
- South Africa (4):
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Department of Medical Oncology, University of Pretoria and Steve Biko, Pretoria, Gauteng
  - Groenkloof Life hospital., Pretoria, Gauteng
  - Department of Haematology, Cape Town, Western Cape
- South Korea (6):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Dong A University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Chonbuk National University Hospital, Jeonju
  - Kangbuk Samsung Hospital, Seoul
  - Seoul St. Mary's Hospital of the Catholic University of Korea, Seoul
- Spain (10):
  - Hospital (Universitari(o)) Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario La Princesa, Madrid, Málaga
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
- Sweden (5):
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Karolinska University Hospital Solna, Stockholm
  - Norrlands University Hospital, Umeå
  - Akademiska Hospital, Uppsala
- Taiwan (4):
  - China Medical University Hospital, Taichung, R.o.c.
  - Chi-Mei Medical Center, Tainan, R.o.c.
  - Mackay Memorial Hospital, Taipei, R.o.c.
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
- Thailand (4):
  - Division of Hematology, Department of Internal Medicine, Maharaj Nakorn Chiang Mai Hospital, Muang, Chiang Mai
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Division of Hematology, Department of Medicine, Faculty of Medicine Siriraj Hospital, Bangkok
- Ukraine (9):
  - MI "Cherkasy Regional Oncological Dispensary " of Cherkasy Regional Council, Cherkasy
  - Regional Clinical Hospital in Ivano-Frankivsk, Hematology Department, Ivano-Frankivsk
  - Khmelnytskyi Regional Hospital, Hematology Department, Khmelnytskyi
  - State Institution "National research center for radiation medicine of NAMS of Ukraine",, Kyiv
  - State Institution "National research center for radiation medicine of NAMS of Ukraine", Kyiv
  - transplantation department of hemotology and transplantology division within Clinical Radiology, Kyiv
  - Chair of internal medicine #2., Kyiv
  - Kyiv City Clinical Hospital #9, Hematology department #1,, Kyiv
  - State Institution "Institute of Blood Pathology and Transfusion Medicine NAMS of Ukraine", Lviv
- United Kingdom (9):
  - Catherine Lewis Centre, Hammersmith Hospital, London, Greater London
  - Linda McCartney Centre, Liverpool, Merseyside
  - Department of Clinical Haematology, Nottingham, Nottinghamshire
  - Cancer & Haematology Centre, Churchill Hospital, Oxford, Oxfordshire
  - Department of Haematology The Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Heartlands Hospital, Birmingham, WEST Midlands
  - St James's Institute of Oncology, Leeds, WEST Yorkshire
  - Department of Haematology, Cardiff
  - The Hope Clinical Trials Facility, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Garrett M, Knight B, Cortes JE, Deininger MW. Population modeling of bosutinib exposure-response in patients with newly diagnosed chronic phase chronic myeloid leukemia. Cancer Med. 2023 Sep;12(17):17981-17992. doi: 10.1002/cam4.6439. Epub 2023 Aug 8. PMID 37553873
- [Derived] Brummendorf TH, Cortes JE, Milojkovic D, Gambacorti-Passerini C, Clark RE, le Coutre P, Garcia-Gutierrez V, Chuah C, Kota V, Lipton JH, Rousselot P, Mauro MJ, Hochhaus A, Hurtado Monroy R, Leip E, Purcell S, Yver A, Viqueira A, Deininger MW; BFORE study investigators. Bosutinib versus imatinib for newly diagnosed chronic phase chronic myeloid leukemia: final results from the BFORE trial. Leukemia. 2022 Jul;36(7):1825-1833. doi: 10.1038/s41375-022-01589-y. Epub 2022 May 28. PMID 35643868
- [Derived] Takahashi N, Cortes JE, Sakaida E, Ishizawa K, Ono T, Doki N, Matsumura I, Garcia-Gutierrez V, Rosti G, Ono C, Ohkura M, Tanetsugu Y, Viqueira A, Brummendorf TH. Safety profile of bosutinib in Japanese versus non-Japanese patients with chronic myeloid leukemia: a pooled analysis. Int J Hematol. 2022 Jun;115(6):838-851. doi: 10.1007/s12185-022-03314-y. Epub 2022 Mar 2. PMID 35235189
- [Derived] Chuah C, Koh LP, Numbenjapon T, Zang DY, Ong KH, Do YR, Ohkura M, Ono C, Viqueira A, Cortes JE, Brummendorf TH. Efficacy and safety of bosutinib versus imatinib for newly diagnosed chronic myeloid leukemia in the Asian subpopulation of the phase 3 BFORE trial. Int J Hematol. 2021 Jul;114(1):65-78. doi: 10.1007/s12185-021-03144-4. Epub 2021 Apr 13. PMID 33851349
- [Derived] Cortes JE, Gambacorti-Passerini C, Deininger MW, Mauro MJ, Chuah C, Kim DW, Dyagil I, Glushko N, Milojkovic D, le Coutre P, Garcia-Gutierrez V, Reilly L, Jeynes-Ellis A, Leip E, Bardy-Bouxin N, Hochhaus A, Brummendorf TH. Bosutinib Versus Imatinib for Newly Diagnosed Chronic Myeloid Leukemia: Results From the Randomized BFORE Trial. J Clin Oncol. 2018 Jan 20;36(3):231-237. doi: 10.1200/JCO.2017.74.7162. Epub 2017 Nov 1. PMID 29091516

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib: Participants with Philadelphia chromosome-positive chronic myeloid leukemia (CML) received bosutinib tablets at a dose of 400 milligram (mg), orally once daily in the core treatment phase of 12 months and continued the same treatment into the extension phase or followed up for safety for up to approximately 4 years, until the end of the study, treatment failure, unacceptable toxicity, death, or withdrawal of consent, whichever occurred first.
- Imatinib: Participants with Philadelphia chromosome-positive CML received imatinib tablets at a dose of 400 mg, orally once daily in the core treatment phase of 12 months and continued the same treatment into the extension phase or followed up for safety for up to approximately 4 years, until the end of the study, treatment failure, unacceptable toxicity, death, or withdrawal of consent, whichever occurred first.
Period: Overall Study
Arm/Group | Bosutinib | Imatinib
Started | 268 | 268
Treated | 268 | 265
mITT Population | 246 | 241
Completed | 232 | 231
Not Completed | 36 | 37
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Investigator Request | 0 | 2
Not completed — Deceased | 14 | 14
Not completed — Lost to Follow-up | 6 | 7
Not completed — Other | 2 | 1
Not completed — Missing | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants with study drug assignments designated according to initial randomization.
Groups:
- Bosutinib: Participants with Philadelphia chromosome-positive CML received bosutinib tablets at a dose of 400 mg, orally once daily in the core treatment phase of 12 months and continued the same treatment into the extension phase or followed up for safety for up to approximately 4 years, until the end of the study, treatment failure, unacceptable toxicity, death, or withdrawal of consent, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Bosutinib | Imatinib | Total
Number analyzed (Participants) | 268 | 268 | 536
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (15.40) | 50.9 (14.43) | 50.9 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 113 | 225
  Male | 156 | 155 | 311

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Molecular Response (MMR) at Month 12
Description: MMR was defined as a ratio of breakpoint cluster region to abelson (BCR-ABL/ABL) less than or equal to (<=) 0.1 percent (%) on the international scale (IS) (greater than or equal to [>=] 3 log reduction from standardized baseline in ratio of BCR-ABL to ABL transcripts [>=3000 ABL required]) by quantitative reverse transcriptase polymerase chain reaction (RT-qPCR). The percentage of participants with MMR at Month 12 are reported.
Time Frame: Month 12
Population: Modified intent-to-treat (mITT) population included all randomized participants with Philadelphia chromosome positive (Ph+) CML harboring the b2a2 and/or b3a2 transcript and baseline BCR-ABL copies greater than (>) 0 with study drug assignment designated according to initial randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 246 | 241
percentage of participants | 47.2 [40.9 to 53.4] | 36.9 [30.8 to 43.0]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; A total sample size of 500 Ph+ participants is required for the study to provide >= 90% power to detect at least 15% difference (assuming 25% in the imatinib vs 40% in the bosutinib arm) in the MMR rates at 12 months (48 weeks) with a 1-sided alpha of 2.5%, and 2 interim futility analyses at 33% and 66% of patients with adequate follow-up with early stopping for futility only (non-binding, O'Brien-Fleming analog beta spending function); Test type: Superiority; p = 0.0100, Cochran-Mantel-Haenszel — 1-sided p-value based on CMH test for general association between treatment and response with stratification by sokal risk group (low, intermediate, high) and region (1-3) at time of randomization. Statistical significance threshold: 1-sided 0.025; Odds Ratio (OR) = 1.547, 95% CI 2-sided [1.072 to 2.233] — 95% Confidence Interval (CI) for the odds ratio adjusted for sokal risk group and region are based on Mantel-Haenszel confidence limits

2. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) Up to Month 18
Description: MMR was defined as a ratio of BCR-ABL/ABL <=0.1% on the international scale (>=3 log reduction from standardized baseline in ratio of BCR-ABL to ABL transcripts [>=3000 ABL required]) by quantitative RT-qPCR. The percentage of participants with MMR for up to Month 18 are reported.
Time Frame: Up to Month 18
Population: mITT population included all randomized participants with Ph+ CML harboring the b2a2 and/or b3a2 transcript and baseline BCR-ABL copies >0 with study drug assignment designated according to initial randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 246 | 241
percentage of participants | 61.0 [54.9 to 67.1] | 52.7 [46.4 to 59.0]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; If the primary analysis was significant, each member of the short-term family (CCyR by Month 12, MMR by Month 18) was tested via Bonferroni's procedure at the 1-sided level of 0.0125; Test type: Superiority; p = 0.0303, Cochran-Mantel-Haenszel — 1-sided p-value based on CMH test for general association between treatment and response with stratification by sokal risk group (low, intermediate, high) and region (1-3) at time of randomization. Statistical significance threshold: 1-sided 0.0125; Odds Ratio (OR) = 1.418, 95% CI 2-sided [0.986 to 2.037] — 95% CI for the odds ratio adjusted for sokal risk group and region are based on Mantel-Haenszel confidence limits

3. Secondary Outcome: Kaplan-Meier Estimate of Probability of Retaining Major Molecular Response (MMR) at Month 48
Description: The Kaplan-Meier curve was generated based on the first date of MMR until the date of the confirmed loss of MMR or censoring, objectively documented, for responders only. Confirmed loss of MMR was BCR-ABL/ABL IS ratio >0.1% in association with a >=5-fold increase in BCR-ABL/ABL IS ratio from the lowest value achieved up to that time-point confirmed by a second assessment at least 28 days later. Treatment discontinuation due to suboptimal response/treatment failure, progressive disease (PD) or death due to PD within 28 days of last dose were considered confirmed loss of MMR. PD was defined as disease progression to accelerated phase (AP) or blast phase (BP) CML.
Time Frame: Month 48
Population: mITT population included all randomized participants with Ph+ CML harboring the b2a2 and/or b3a2 transcript and baseline BCR-ABL copies >0 with study drug assignment designated according to initial randomization and who achieved MMR (responders). Here, "Overall number of Participants Analyzed (N)" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 182 | 158
percentage of participants | 92.2 [86.8 to 95.4] | 92.0 [85.9 to 95.5]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; The medians have not been reached in either arm, as such, the premature estimated hazard ratio is provided; Test type: Superiority; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.49 to 2.44] — Hazard ratio (95% CIs) are based on the treatment effect (Bosutinib compared with Imatinib) in a stratified (by Sokal risk group at randomization and region) Cox proportional hazards model for the hazard of the respective event

4. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR) Up to Month 12
Description: Complete Cytogenetic Response (CCyR) was based on the prevalence of Ph+ metaphases among cells in metaphase on a bone marrow (BM) aspirate. CCyR was achieved when there was 0% Ph+ metaphases among cells in a BM sample when at least 20 metaphases from a BM sample were analyzed, or MMR if no BM was available. The percentage of participants with CCyR for up to Month 12 are reported.
Time Frame: Up to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 246 | 241
percentage of participants | 77.2 [72.0 to 82.5] | 66.4 [60.4 to 72.4]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0037, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.740, 95% CI 2-sided [1.160 to 2.610] — 95% CI for the odds ratio adjusted for sokal risk group and region are based on Mantel-Haenszel confidence limits

5. Secondary Outcome: Kaplan-Meier Estimate of Probability of Retaining Complete Cytogenetic Response (CCyR) at Month 48
Description: The Kaplan-Meier curve was generated based on the first date of CCyR until the date of the confirmed loss of CCyR or censoring, objectively documented, for responders only. Confirmed loss of CCyR was the presence of at least one Ph+ metaphase confirmed by a second assessment at least 28 days later. Treatment discontinuation due to suboptimal response/treatment failure, PD or death due to PD within 28 days of last dose were considered confirmed loss of CCyR. PD was defined as disease progression to AP or BP CML.
Time Frame: Month 48
Population: mITT population included all randomized participants with Ph+ CML harboring the b2a2 and/or b3a2 transcript and baseline BCR-ABL copies >0 with study drug assignment designated according to initial randomization and who achieved CCyR (responders). Here, "N" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 205 | 185
percentage of participants | 97.4 [93.9 to 98.9] | 93.7 [88.9 to 96.5]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; The medians have not been reached in either arm, as such, the premature estimated hazard ratio is provided; Test type: Superiority; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.14 to 1.13] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Cumulative Incidence of Event Free Survival (EFS) Events
Description: EFS was defined as time from randomization to death due to any cause, transformation to AP or BP at any time, confirmed loss of complete hematologic response (CHR), confirmed loss of CCyR or censoring. Loss of CHR was defined as a hematologic assessment of non-CHR (chronic phase, AP, or BP) confirmed by 2 assessments at least 4 weeks apart. Loss of CHR was defined as appearance of any of the following: WBC count that rises to >20.0*10^9/L, platelet count rises to >=600*10^9/L, appearance of palpable spleen or other extramedullary involvement proven by biopsy, appearance of 5% myelocytes in peripheral blood, appearance of blasts or promyelocytes in peripheral blood. Loss of CCyR was defined as at least 1 Ph+ metaphase from analysis of <100 metaphases confirmed by follow up cytogenetic analysis after 1 month. Cumulative incidence of EFS was defined as percentage of participants with EFS event at Month 60 and was adjusted for competing risk of treatment discontinuation without event.
Time Frame: Up to Month 60
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 246 | 241
percentage of participants | 6.9 [4.2 to 10.5] | 10.4 [6.9 to 14.6]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; If each member of the short-term family (CCyR by Month 12, MMR by Month 18) was significant, EFS and OS were tested sequentially via the Holm's testing procedure at the 1-sided family wise level of 0.025. If one member of the short-term family was significant, EFS and OS were tested sequentially at 1-sided 0.0125; Test type: Superiority; p = 0.0749, Gray's test — 1-sided p-value based on Gray's test for comparing cumulative incidence function between treatment arms stratified by sokal risk group (low, intermediate, high) and region (1-3). Statistical significance threshold: 1-sided 0.0125; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.35 to 1.17] — The hazard ratio (95% CIs) are based on the proportional subdistribution hazards model stratified by Sokal risk group and region

7. Secondary Outcome: Overall Survival (OS) Rate
Description: OS was defined as the time (in months) from randomization to the occurrence of death due to any cause or censoring. Kaplan-meier analysis was used for determination of OS. Percentage of participants who were alive were estimated in this outcome measure.
Time Frame: Up to Month 60
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 246 | 241
percentage of participants | 94.9 [91.1 to 97.0] | 94.0 [90.1 to 96.4]
Statistical Analysis 1: Comparison: Bosutinib vs Imatinib; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.2827, Log Rank — 1-sided p-value based on log-rank test for comparing survival curves between treatment arms stratified by sokal risk group and region. OS was not tested as EFS was not significant; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.37 to 1.73] — The hazard ratio (95% CIs) are based on the treatment effect (Bosutinib compared with Imatinib) in a stratified (by Sokal risk group at randomization and region) Cox proportional hazards model for the hazard of the respective event

8. Other Pre Specified Outcome: Summary of Trough Plasma Concentration by Complete Cytogenetic Response (CCyR) of Bosutinib
Description: CCyR was based on the prevalence of Ph+ metaphases among cells in metaphase on a BM aspirate. CCyR was achieved when there was 0% Ph+ metaphases among cells in a BM sample when at least 20 metaphases from a BM sample were analyzed, or MMR if no BM was available. Trough plasma concentration of participants who had CCyR are presented in this outcome measure.
Time Frame: Pre-dose on Days 28, 56 and 84
Population: Pharmacokinetic (PK) population included all enrolled participants who received at least 1 dose of bosutinib and had sufficient plasma results available. Here, "N" signifies number of participants evaluable for this outcome measure and "number analyzed (n)" signifies participants evaluable at specified time points only. Data for this outcome measure was not planned to be collected and analyzed for Imatinib arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Bosutinib
Number analyzed (Participants) | 191
nanogram per milliliter (ng/mL)
  Day 28: number analyzed (Participants) | 181
  Day 28 | 71.282 (46.0545)
  Day 56: number analyzed (Participants) | 184
  Day 56 | 73.069 (45.1349)
  Day 84: number analyzed (Participants) | 184
  Day 84 | 83.973 (64.3206)

9. Other Pre Specified Outcome: Summary of Trough Plasma Concentration by Major Molecular Response (MMR) of Bosutinib
Description: MMR was defined as a ratio of BCR-ABL/ABL <=0.1% on the international scale (>=3 log reduction from standardized baseline in ratio of BCR-ABL to ABL transcripts) by quantitative RT-qPCR. Trough plasma concentration of participants who had MMR are presented in this outcome measure.
Time Frame: Pre-dose on Days 28, 56 and 84
Population: PK population included all enrolled participants who received at least 1 dose of bosutinib and had sufficient plasma results available. Here, "N" signifies number of participants evaluable for this outcome measure and "n" signifies participants evaluable at specified time points only. Data for this outcome measure was not planned to be collected and analyzed for Imatinib arm as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 141
ng/mL
  Day 28: number analyzed (Participants) | 140
  Day 28 | 75.050 (51.9551)
  Day 56: number analyzed (Participants) | 140
  Day 56 | 78.437 (43.6019)
  Day 84 | 91.081 (72.1500)

10. Other Pre Specified Outcome: Summary of Trough Plasma Concentration by Presence of Grade 1 or Higher Adverse Events (AEs) of Bosutinib
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to maximum severity grading based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 1= mild; Grade 2= moderate; within normal limits, Grade 3= severe or medically significant but not immediately life-threatening; Grade 4= life-threatening or disabling; urgent intervention indicated; Grade 5= death. Trough plasma concentration of participants who had grade 1 or higher AE are presented in this outcome measure. Data of plasma concentration is reported separately for each preferred term of AE.
Time Frame: Pre-dose on Days 28, 56 and 84
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 177
ng/mL
  Day 28: Diarrhea | 69.402 (55.5005)
  Day 28: Thrombocytopenia: number analyzed (Participants) | 60
  Day 28: Thrombocytopenia | 63.529 (40.9949)
  Day 28: Rash: number analyzed (Participants) | 84
  Day 28: Rash | 74.779 (60.6257)
  Day 28: Nausea: number analyzed (Participants) | 86
  Day 28: Nausea | 66.011 (42.6437)
  Day 28: Vomiting: number analyzed (Participants) | 44
  Day 28: Vomiting | 71.684 (60.7208)
  Day 56: Diarrhea: number analyzed (Participants) | 172
  Day 56: Diarrhea | 68.834 (42.6621)
  Day 56: Thrombocytopenia: number analyzed (Participants) | 61
  Day 56: Thrombocytopenia | 65.327 (43.2859)
  Day 56: Rash: number analyzed (Participants) | 84
  Day 56: Rash | 70.016 (38.7506)
  Day 56: Nausea: number analyzed (Participants) | 85
  Day 56: Nausea | 61.626 (44.4007)
  Day 56: Vomiting: number analyzed (Participants) | 40
  Day 56: Vomiting | 65.980 (45.9064)
  Day 84: Diarrhea: number analyzed (Participants) | 165
  Day 84: Diarrhea | 81.269 (64.6462)
  Day 84: Thrombocytopenia: number analyzed (Participants) | 63
  Day 84: Thrombocytopenia | 71.585 (33.6674)
  Day 84: Rash: number analyzed (Participants) | 85
  Day 84: Rash | 89.080 (69.5237)
  Day 84: Nausea: number analyzed (Participants) | 80
  Day 84: Nausea | 77.702 (61.6179)
  Day 84: Vomiting: number analyzed (Participants) | 41
  Day 84: Vomiting | 86.949 (55.3041)

11. Other Pre Specified Outcome: Summary of Trough Plasma Concentration by Presence of Grade 3 or Higher Adverse Events (AEs) of Bosutinib
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to maximum severity grading based on NCI CTCAE version 4.0. Grade 1= mild; Grade 2= moderate; within normal limits, Grade 3= severe or medically significant but not immediately life-threatening; Grade 4= life-threatening or disabling; urgent intervention indicated; Grade 5= death. Trough plasma concentration of participants who had grade 3 or higher AE are presented in this outcome measure. Data of plasma concentration is reported separately for each preferred term of AE.
Time Frame: Pre-dose on Days 28, 56 and 84
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 24
ng/mL
  Day 28: Diarrhea: number analyzed (Participants) | 19
  Day 28: Diarrhea | 87.769 (102.6181)
  Day 28: Thrombocytopenia: number analyzed (Participants) | 23
  Day 28: Thrombocytopenia | 49.220 (36.3461)
  Day 28: Rash: number analyzed (Participants) | 4
  Day 28: Rash | 71.150 (43.3246)
  Day 28: Vomiting: number analyzed (Participants) | 3
  Day 28: Vomiting | 14.663 (21.5799)
  Day 56: Diarrhea: number analyzed (Participants) | 16
  Day 56: Diarrhea | 68.513 (45.2672)
  Day 56: Thrombocytopenia | 56.853 (34.3892)
  Day 56: Rash: number analyzed (Participants) | 4
  Day 56: Rash | 58.925 (18.8656)
  Day 56: Vomiting: number analyzed (Participants) | 1
  Day 56: Vomiting | 38.200 (NA) — As only 1 participant was analyzed, standard deviation could not be calculated.
  Day 84: Diarrhea: number analyzed (Participants) | 17
  Day 84: Diarrhea | 76.782 (46.3006)
  Day 84: Thrombocytopenia: number analyzed (Participants) | 23
  Day 84: Thrombocytopenia | 67.623 (35.3084)
  Day 84: Rash: number analyzed (Participants) | 3
  Day 84: Rash | 83.967 (19.2542)
  Day 84: Vomiting: number analyzed (Participants) | 1
  Day 84: Vomiting | 12.400 (NA) — As only 1 participant was analyzed, standard deviation could not be calculated.

12. Other Pre Specified Outcome: Number of Participants With Vital Signs Abnormalities
Description: Criteria for vital signs abnormalities: systolic blood pressure <80 millimeter of mercury (mmHg), >210 mmHg; diastolic blood pressure <40 mmHg, >130 mmHg; heart rate <40 beats per minute (bpm), >150 bpm; temperature <32 degree celsius, >40 degree celsius; weight >=10% increase from baseline, >=10% decrease from baseline. The number of participants with any vital sign abnormalities during On-treatment period are reported. On-Treatment was defined as values collected after the date of the first dose of test article until the last date of test article +28 days.
Time Frame: Baseline up to end of treatment (up to Month 60)
Population: Safety population included all participants who received at least 1 dose of study medication with treatment assignments designated to actual study treatment received. Here, "N" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 262 | 263
Participants | 107 | 109

13. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities Based on National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) Version 4.03
Description: Laboratory parameters included hematological (haemoglobin, lymphocytes [absolute], neutrophils [absolute], platelets and leukocytes) and biochemistry (albumin, alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, amylase, bilirubin, creatinine kinase, calcium, creatinine, glucose, potassium, lipase, magnesium, phosphate, sodium, urate) parameters. Abnormalities in laboratory tests were graded by NCI CTCAE version 4.03 as Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. The number of participants with laboratory test abnormalities were reported.
Time Frame: Baseline up to end of treatment (up to Month 60)
Population: Safety population included all participants who received at least 1 dose of study medication with treatment assignments designated to actual study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 268 | 265
Participants
  Grade 1 | 6 | 7
  Grade 2 | 67 | 59
  Grade 3 | 133 | 154
  Grade 4 | 61 | 45

14. Other Pre Specified Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities included heart rate: increase of >15 bpm from baseline value and >=120 bpm, decrease of >15 bpm from baseline value and <=45 bpm; PR interval: change of >=20 msec from baseline value and >=220 milliseconds (msec); QRS interval >=120 msec; QTcB interval >500 msec, increase of >60 msec from baseline; >450 msec (Men) or >470 msec (Women). QT interval using Fridericia's correction (QTcF) >500 msec, increase of >60 msec from baseline, >450 msec (Men) or >470 msec (Women). The number of participants with ECG abnormalities during On-treatment period are reported. On-Treatment was defined as values collected after the date of the first dose of test article up until the last date of test article +28 days.
Time Frame: Baseline up to end of treatment (up to Month 60)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 266 | 262
Participants | 16 | 13

15. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) Leading to Study Drug Discontinuation
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to end of treatment (up to Month 60)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 268 | 265
Participants | 68 | 38

16. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events by National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 4.0)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity grading based on NCI CTCAE version 4.0. Grade 1 =mild; Grade 2 =moderate; Grade 3 =severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; Grade 4 =life-threatening or disabling, urgent intervention indicated; Grade 5 =death. Treatment-emergent events were events between first dose of study drug and up to 60 months that were absent before treatment that worsened relative to pretreatment state. If the same participant in a given treatment had more than 1 adverse event, only the maximum CTCAE was reported.
Time Frame: Baseline up to end of treatment (up to Month 60)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib | Imatinib
Number analyzed (Participants) | 268 | 265
Participants
  Grade 1 | 7 | 24
  Grade 2 | 61 | 86
  Grade 3 | 144 | 120
  Grade 4 | 50 | 28
  Grade 5 | 3 | 4

ADVERSE EVENTS:
Time Frame: From first dose of drug up to 28 days after last dose (up to Month 60)
Description: All-cause mortality: The total number of deaths occurred during study (from randomization and up to month 60) are reported for all randomized participants, not only for treated participants, and included deaths which occurred after 28 days post last study drug dose. Serious AEs and other AEs: Analysis performed on safety population. The safety population included all participants, regardless of Philadelphia chromosome or transcript status, who received at least 1 dose of study medication.
Arm/Group | Bosutinib | Imatinib
All-Cause Mortality (participants affected / at risk) | 14/268 | 14/268
Serious Adverse Events (participants affected / at risk) | 98/268 | 68/265
Other Adverse Events (participants affected / at risk) | 264/268 | 260/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=268) | Imatinib (N=265)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 4 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Thyroid disorder (Endocrine disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Necrotising oesophagitis (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 1
General physical health deterioration (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Implant site haematoma (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Swelling face (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 5
Gastroenteritis (Infections and infestations) | 6 | 1
Cellulitis (Infections and infestations) | 3 | 2
Influenza (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Abscess (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 2
Appendicitis perforated (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Candida pneumonia (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Fournier's gangrene (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1
Infective pericardial effusion (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Meningococcal sepsis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Oropharyngitis fungal (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Splenic infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 6 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fallopian tube cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Prostatic dysplasia (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Pregnancy of partner (Social circumstances) | 2 | 1
Embolism (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=268) | Imatinib (N=265)
Thrombocytopenia (Blood and lymphatic system disorders) | 96 | 53
Anaemia (Blood and lymphatic system disorders) | 59 | 59
Neutropenia (Blood and lymphatic system disorders) | 33 | 61
Leukopenia (Blood and lymphatic system disorders) | 18 | 34
Lymphopenia (Blood and lymphatic system disorders) | 15 | 8
Periorbital oedema (Eye disorders) | 4 | 44
Eyelid oedema (Eye disorders) | 3 | 24
Conjunctival haemorrhage (Eye disorders) | 2 | 18
Dry eye (Eye disorders) | 4 | 16
Lacrimation increased (Eye disorders) | 1 | 18
Vision blurred (Eye disorders) | 5 | 14
Diarrhoea (Gastrointestinal disorders) | 201 | 106
Nausea (Gastrointestinal disorders) | 100 | 112
Vomiting (Gastrointestinal disorders) | 55 | 54
Abdominal pain (Gastrointestinal disorders) | 61 | 25
Abdominal pain upper (Gastrointestinal disorders) | 28 | 26
Constipation (Gastrointestinal disorders) | 36 | 17
Dyspepsia (Gastrointestinal disorders) | 26 | 24
Abdominal distension (Gastrointestinal disorders) | 14 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 14
Toothache (Gastrointestinal disorders) | 14 | 7
Fatigue (General disorders) | 57 | 54
Pyrexia (General disorders) | 44 | 29
Oedema peripheral (General disorders) | 20 | 43
Asthenia (General disorders) | 34 | 24
Face oedema (General disorders) | 7 | 17
Influenza like illness (General disorders) | 16 | 6
Upper respiratory tract infection (Infections and infestations) | 36 | 33
Nasopharyngitis (Infections and infestations) | 36 | 30
Urinary tract infection (Infections and infestations) | 26 | 18
Influenza (Infections and infestations) | 24 | 14
Gastroenteritis (Infections and infestations) | 12 | 17
Bronchitis (Infections and infestations) | 19 | 6
Sinusitis (Infections and infestations) | 15 | 8
Alanine aminotransferase increased (Investigations) | 90 | 16
Aspartate aminotransferase increased (Investigations) | 69 | 18
Lipase increased (Investigations) | 56 | 30
Blood creatine phosphokinase increased (Investigations) | 14 | 33
Blood creatinine increased (Investigations) | 18 | 22
Amylase increased (Investigations) | 25 | 10
Weight increased (Investigations) | 8 | 20
Blood alkaline phosphatase increased (Investigations) | 17 | 7
Blood bilirubin increased (Investigations) | 17 | 7
Decreased appetite (Metabolism and nutrition disorders) | 29 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 23
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 | 49
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 81
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 39
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 48
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 19
Headache (Nervous system disorders) | 58 | 41
Dizziness (Nervous system disorders) | 25 | 23
Insomnia (Psychiatric disorders) | 18 | 19
Anxiety (Psychiatric disorders) | 15 | 15
Depression (Psychiatric disorders) | 9 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 10
Rash (Skin and subcutaneous tissue disorders) | 61 | 39
Pruritus (Skin and subcutaneous tissue disorders) | 30 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 16
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 14
Hypertension (Vascular disorders) | 26 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.